CLINICAL TRIAL: NCT04105361
Title: Impact of Posterior Nasal Neurectomy With Functional Endoscopic Sinus Surgery for Chronic Rhinosinusitis With Nasal Polyposis :A Comparative Study
Brief Title: Impact of Posterior Nasal Neurectomy With Functional Endoscopic Sinus Surgery for Chronic Rhinosinusitis With Nasal Polyposis:A Comparative Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ET Zarief, Principle investigator, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Nasal polyposis
Record Dates: First submitted 2019-09-25; First posted 2019-09-26 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Nasal Polyps
MeSH Terms: conditions — Nasal Polyps

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): We will do posterior nasal neurectomy in patients with allergic rhinitis after FESS in one side of the nose
  Interventions: Procedure: Posterior neurectomy
- Control group (Experimental): We will do FESS only in the other side of the nose
  Interventions: Procedure: Posterior neurectomy

INTERVENTIONS:
Procedure: Posterior neurectomy — Cut of posterior nasal nerve

SUMMARY:
The study will be conducted to investigate the efficacy of posterior nasal neurectomy in control of recurrence and improvment of allergic symptoms in patients with allergic rhinitis combined with nasal polyposis

DETAILED DESCRIPTION:
Allergic rhinitis patients with nasal polyposis will go through FESS combined with posterior nasal neurectomy to detect recurrence rate

ELIGIBILITY:
Inclusion Criteria:

* all cases presented to ENT department Assuit University with allergic rhinosinusitis with nasal polyposis

Exclusion Criteria:

* refusing enrollment into the study. Pregnant women Refusing surgery Containdication to surgery Patients with aspirin syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Impact of posterior nasal neurectomy on recurrence rate in allergic rhinosinusitis with nasal polyposis | 1 year
  Surgical procedure to evaluate the recurrence of nasal polyposis

REFERENCES:
- [Background] Mengeling WL. Anamnestic immune response of pigs to pseudorabies virus: latent virus reactivation versus direct oronasal and parenteral exposure to virus. J Vet Diagn Invest. 1991 Apr;3(2):133-6. doi: 10.1177/104063879100300205. PMID 1654132